CLINICAL TRIAL: NCT06301269
Title: A Study on Self-Compassion,Depression,and Quality of Life Among Primary Caregivers of People With Dementia
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202312124RINA
Record Dates: First submitted 2024-03-03; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Dementia
Keywords: dementia; self-compassion; Primary Caregivers
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
The goal of this observational study is to investigate the correlation between self-compassion, depression, and quality of life among primary caregivers of persons with dementia.

The main questions it aims to answer are:

1. What is the current status of self-compassion, depression, and quality of life among primary caregivers of persons with dementia?
2. Are there differences in self-compassion, depression, and quality of life among primary caregivers of persons with dementia based on different background variables?
3. What is the correlation between self-compassion, depression, and quality of life among primary caregivers of persons with dementia?

Participants will fill out the questionnaire to complete the study.

DETAILED DESCRIPTION:
The study design of this research is cross-sectional. The participants are primary caregivers of dementia patients diagnosed by specialists, aged 18 and above, who spend 8 hours or more daily (including overnight caregivers) providing care. Data is collected using instruments including the Self-Compassion Scale, the PHQ-9 Scale (Patient Health Questionnaire,PHQ-9）, and the Quality-of-Life Scale to investigate the relationship between self-compassion, depression, and quality of life among primary caregivers of dementia patients.

The study uses independent samples t-tests and one-way ANOVA( analysis of variance,ANOVA) to explore differences in self-compassion, depression, and quality of life among primary caregivers of dementia patients based on different background variables. Pearson correlation is used to analyze the relationships between these variables. Finally, linear regression is used to predict the performance of primary caregivers of dementia patients in self-compassion, depression, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. primary caregivers of dementia patients diagnosed by specialists
2. aged 18 and above
3. who spend 8 hours or more daily (including overnight caregivers) providing care

Exclusion Criteria:

1. Those who do not agree to participate in the research
2. Caregivers in a paid relationship with dementia patients, such as foreign domestic helpers and government-provided resident care attendant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will include primary caregivers of people with dementia. Participants will be adults aged 18 years and older who are currently providing care for a family member , Participants will be recruited from NTUH Neurology ward and Out-Patient Departments (OPD).
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-03-10 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Self-Compassion Scale | The participants will spend 5-10 minutes completing the questionnaire during the study
  The self-compassion score, measured using the Self-Compassion Scale, reflects the level of self-compassion among primary caregivers of people with dementia.
PHQ-9 Scale | The participants will spend 5-10 minutes completing the questionnaire during the study
  The PHQ-9 Scale, measured using the PHQ-9 Scale, reflects the level of depression among primary caregivers of people with dementia.
Quality-of-Life Scale | The participants will spend 5-10 minutes completing the questionnaire during the study
  The Quality-of-Life Scale , measured using the Quality-of-Life Scale , reflects the level of Quality-of-Life among primary caregivers of people with dementia.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan